CLINICAL TRIAL: NCT01259817
Title: Single Arm Salvage Therapy With Pegylated Interferon Alfa-2a for Patients With High Risk Polycythemia Vera or High Risk Essential Thrombocythemia Who Are Either Hydroxyurea Resistant or Intolerant or Have Had Abdominal Vein Thrombosis
Brief Title: Pegylated Interferon Alfa-2a Salvage Therapy in High Risk Polycythemia Vera (PV) or Essential Thrombocythemia (ET)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ronald Hoffman (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH); Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Ronald Hoffman, Professor of Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 09-1300 001; P01CA108671 (NIH); MPD-RC 111 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2010-12-06; First posted 2010-12-14 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: High Risk Polycythemia Vera; High Risk Essential Thrombocythemia
Keywords: Polycythemia Vera; Essential Thrombocythemia; Hydroxyurea Resistant; Abdominal Vein Thrombosis; PEGASYS
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential | interventions — peginterferon alfa-2a; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEGASYS (Experimental): Patient will start at 45 micrograms per week and gradually increase to 180 micrograms per week. Pegasys will be supplied in prefilled syringes and are to be given subcutaneously.
  Interventions: Drug: PEGASYS
- Aspirin (Active Comparator): 81 or 100 mg daily.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: PEGASYS — Patient will start at 45 micrograms per week and gradually increase to 180 micrograms per week. Pegasys will be supplied in prefilled syringes and are to be given subcutaneously.
  Other Names: Pegylated Interferon Alfa-2a
  Arms: PEGASYS
Drug: Aspirin — 81 or 100 mg daily.
  Other Names: acetylsalicylic acid
  Arms: Aspirin

SUMMARY:
The aim of this research is to look at two conditions, Essential Thrombocythemia (ET) and Polycythemia Vera (PV). ET causes people to produce too many blood cells called platelets and PV causes too many platelets and red blood cells to be made. Platelets are particles which circulate in the blood stream and normally prevent bleeding and bruising. Having too many platelets in the blood increases the risk of developing blood clots, which can result in life threatening events like heart attacks and strokes. When the number of red blood cells is increased in PV this will slow the speed of blood flow in the body and increases the risk of developing blood clots.

It is important for patients with ET or PV who are at risk of blood clots to receive drugs which will minimize the risks of developing these blood clots but at the moment the investigators are not sure which drugs will best control the disorder.

The purpose of this study is to look at the effectiveness of giving patients who have been diagnosed with ET and PV a study drug regimen using Aspirin and PEGASYS (also known as Pegylated interferon alfa-2a, instead of the standard treatment drug called Hydroxyurea (or hydroxycarbamide or Hydroxyurea), for whom this drug may not be suitable. The drug may not be suitable either because it is not adequately controlling the number of blood cells or some specific side effects occur.

DETAILED DESCRIPTION:
Myeloproliferative disorders (MPDs) are clonal hematologic diseases characterized by the excess production of one or more lineages of mature blood cells, a predisposition to bleeding and thrombotic complications, extramedullary hematopoiesis, and a variable progression to acute leukemia. The classical Philadelphia chromosome-negative MPDs are polycythemia vera (PV), characterized by an expansion in red blood cell production; essential thrombocythemia (ET), characterized by an isolated elevation in the platelet count; and myelofibrosis, distinguished by a fibrotic bone marrow and peripheral blood cytopenias, and accompanied by the highest risk of leukemic transformation. Myelofibrosis can arise de novo, as primary myelofibrosis (PMF), or can evolve out of PV or ET as those diseases progress (so called post-PV MF and post-ET MF). Amongst the MPDs, those characterized by myelofibrosis (PMF together with post-PV and post-ET MF) carry the worst prognosis, with a median survival on the order of 3 to 5 years. Patients typically present with anemia, often requiring transfusions, symptomatic splenomegaly and severe constitutional symptoms. Donor stem cell transplantation is the only potentially curative therapy. To date there is no therapy for myelofibrosis that has been shown to offer a survival benefit, and all other therapies for myelofibrosis are palliative.

In 2005, a major breakthrough in understanding the pathophysiology of MPDs came when 4 groups described a recurrent somatic mutation in Janus kinase 2 (JAK2) in the majority of patients with MPDs. The point mutation in JAK2 encodes a valine to phenylalanine change at position 617 (JAK2 V617F), and confers constitutive tyrosine kinase activity. Introducing the mutation into the bone marrow of mouse models recapitulates the PV phenotype (complete with evolution to bone marrow fibrosis) and inhibitors of JAK2 attenuate the growth of cell lines bearing the mutation in vitro and in vivo, suggesting that JAK2 V617F is a pathophysiologically relevant therapeutic target. It is estimated that 95% of PV cases carry JAK2 V617F, while 50 to 60% of ET and PMF cases are JAK2 V617F+. The discovery of the JAK2V617F mutation in nearly all patients with PV and half those with ET and PMF have redefined the classification and possibly the management of MPNs.

Despite the discovery of the JAK2V617F mutation, many of the clinical questions in the management of MPNs remain unanswered. In PV, for example, cardiovascular mortality remains 1.4 to 1.6 times that of the reference normal population with leukemia and myelofibrosis rates many times increased over baseline. Debate continues over the role of venesection versus cytoreduction as first-line therapy, and whether hydroxycarbamide (Hydroxyurea) is associated with better thrombotic prophylaxis and/or a higher rate of leukemic transformation. Interferons may produce molecular responses in PV patients. In high-risk ET, while Hydroxyurea and aspirin appear to be more optimal than anagrelide and aspirin, vascular complications remain the most significant cause of mortality and morbidity, suggesting that targeting vascular risk factors may be worthwhile.

Furthermore while Hydroxyurea is regarded as the first-choice therapy in most of high risk patients with ET and PV; up to 10% of the patients do not attain the desired reduction of platelet number or hematocrit with the recommended dose of the drug, exhibiting clinical resistance, whereas some will develop unacceptable side effects, demonstrating clinical intolerance.

Quantitation of the JAK2V617F allele burden provides for the first time the opportunity to monitor the effect of potential therapeutic agents on the malignant clone in patients with PV. Great enthusiasm has been expressed for the use of small molecule inhibitors of JAK2 for the treatment of patients with MPN. Phase 1/2 trials have indicated greater than expected toxicity, non specificity of action and an inability of these compounds to dramatically alter the JAK2V617F allele burden. Interferon (rIFN -2b), is a drug that appears to be non-leukemogenic (contrary to 32P, alkylating agents, and possibly Hydroxyurea), and may have a preferential activity on the malignant clone in PV, as suggested by cytogenetic remissions obtained in patients treated with rIFN -2b.

This trial was designed as open-label phase 2 study conducted in two strata of patients with high risk PV or ET who were intolerant of hydroxyurea. Patients with ET or PV with Splanchnic Vein Thrombosis (regardless of prior hydroxyurea) are enrolled in separate strata.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of ET or PV shall be made in accordance with the WHO (2008) criteria (Swerdlow 2008) as shown below (Values below are at the time of diagnosis, not study entry):

* Polycythemia Vera (2 major criteria required)

  1. Hb >18.5g/dl (♂) or 16.5g/dl (♀) or HCT >99 percentile reference range or Elevated red cell mass (>25% above mean predicted value) or Hb >17g/dl (♂) or 15g/dl (♀) if associated with a sustained rise from baseline with no apparent cause (e.g. treated iron deficiency).
  2. Presence of JAK2V617F

     * If source documentation of diagnostic criterion #1 cannot be obtained, then diagnosis can be made with (1) the addition of an erythropoietin level below the reference range of normal AND (2) bone marrow biopsy showing hypercellularity for age with trilineage (panmyelosis) with prominent erythroid, granulocytic, and megakaryocytic proliferation.
* Essential Thrombocythemia (all 6 criteria required)

  1. Platelets count ≥ 450 x 10 to 9/L
  2. Megakaryocyte proliferation with large and mature morphology. No or little granulocyte or erythroid proliferation. Patients may have up to and including 2+ marrow reticulin fibrosis.
  3. Not meeting WHO criteria for CML, PV, MDS, PMF or over myeloid neoplasm
  4. Demonstration of clonal cytogenetic marker or no evidence for a reactive thrombocytosis.
  5. Absence of a leukoerythroblastic blood picture.
  6. May participate in study without presence of JAK2V617F.
* Patients must have high risk disease as defined below:

High risk PV ANY ONE of the following:

* Age ≥ 60 years
* Previous documented thrombosis, erythromelalgia or migraine (severe, recurrent, requiring medications, and felt to be secondary to the MPN) either after diagnosis or within 10 years before diagnosis and considered to be disease related
* Significant (i.e. ≥ 5cm below costal margin on palpation) or symptomatic splenomegaly (splenic infarcts or requiring analgesia)
* Platelets ≥ 1000 x 10 to 9/L
* Diabetes or hypertension requiring pharmacological therapy for ≥ 6 months

High risk ET ANY ONE of the following:

* Age ≥ 60 years
* Platelet count ≥ 1500 x 10 to 9/L
* Previous documented thrombosis, erythromelalgia or migraine (severe, recurrent, requiring medications, and felt to be secondary to the MPN) either after diagnosis or within 10 years before diagnosis and considered to be disease related
* Previous hemorrhage related to ET
* Diabetes or hypertension requiring pharmacological therapy for ≥ 6 months

In addition patients must EITHER be intolerant or resistant to Hydroxyurea according to established criteria as follows:

Any ONE of the following:

* Platelet count ≥ 600 x 10 to 9/L after 3 months of at least 2 g/day of Hydroxyurea (2.5 g/day in patients with a body weight>80 kg)
* WBC < 2.5 x 109/L or Hgb < 11g/dl at any dose of hydroxyurea not to exceed 2g/day.
* Progressive splenomegaly or hepatomegaly (> 5cm from initiation of hydroxyurea) or the appearance of new splenomegaly or hepatomegaly while on MTD of hydroxyurea.
* Not achieving a Hct < 45% in order to eliminate the need for supplemental phlebotomies after 3 months of at least 2g/day or MTD of hydroxyurea.
* Not achieving a WBC of < 10 x 109/L after 3 months of at least 2g/day or MTD of hydroxyurea.
* Having a platelet count < 100 x 109/L on hydroxyurea at any dose without eliminating the need for supplemental phlebotomy or having progressive splenomegaly as defined above.
* Development of a major thrombotic episode (CVA, myocardial infarction, severe migraines requiring medication, abdominal vein thrombosis, deep vein thrombosis) while being treated with maximal tolerated doses of hydroxyurea.
* Presence of leg ulcers or other unacceptable Hydroxyurea-related non-hematological toxicities, such as unacceptable mucocutaneous manifestations, gastrointestinal symptoms, pneumonitis or fever at any dose of Hydroxyurea.

OR have Splanchnic Vein Thrombosis (SVT) (includes Budd-Chiari, abdominal vein thrombosis, portal vein thrombosis, splenic vein thrombosis). For these patients the following additional inclusion/exclusion criteria apply:

* > 3 months since onset of SVT
* SVT treated with oral anticoagulants but no aspirin
* Liver enzymes not > 2 times the normal value
* Absence of encephalopathy, refractory or infected ascites, esophageal varicose of grade > 1 at time of trial entry
* Bone marrow biopsy confirmed diagnosis of PV or ET
* JAK2-V617F mutations present
* These patients may have a normal blood count at trial entry
* Age over 18 years (no upper age limit)
* Able and willing to comply with study criteria
* Signed and informed consent to participant in this study
* Willing to participate in associated correlative science biomarker study
* Serum creatinine < 1.5 x upper limit of normal
* AST and ALT < 2 x upper limit of normal
* Total bilirubin within normal limits

Exclusion Criteria:

* Patients cannot have any other form of chemotherapy for their MPD (other than hydroxyurea). Specifically prior interferon or JAK2 inhibitors are prohibited.
* If a patient has received prior hydroxyurea, they should be tapered off hydroxyurea over a period of the first 2 months of Pegylated interferon alfa-2a therapy. Taper is at the treating physician's discretion, but must be absent (completed) by the start of the third month.
* Patients with a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
* Presence of any life-threatening co-morbidity
* History of active substance or alcohol abuse within the last year
* Any contraindications to pegylated or non-pegylated interferon
* Subjects who have a positive pregnancy test, are pregnant, lactating or of reproductive potential and not practicing an effective means of contraception
* History of psychiatric disorder (e.g. depression; suicidal ideation; psychosis) Subjects with a history of mild depression may be considered for entry into this study, provided that a pretreatment assessment of the subject's affective status supports that the subject is clinically stable based on the investigator's normal practice for such subject.
* History of autoimmune disorder (e.g. hepatitis; ITP; scleroderma; severe psoriasis affecting > 10% of the body, rheumatoid arthritis requiring more than intermittent NSAID for management)
* Hypersensitivity to IFN-α
* HBV or untreated systemic infection
* Known HIV disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration) or clinically relevant ophthalmological disorder (e.g. due to diabetes mellitus or hypertension)
* History or other evidence of decompensated liver disease
* History or other evidence of chronic pulmonary disease associated with functional limitation
* Thyroid dysfunction not adequately controlled
* Any investigational drug <6 weeks prior to the first dose of study drug or not recovered from effects of prior investigational agent.
* Presence of JAK2 exon 12 mutation
* Patients should not meet criteria for post PV or post ET-MF (see appendix B)
* Previous exposure to any formulation of interferon
* Subjects with any other medical condition, which in the opinion of the investigator would compromise the results of the study by deleterious effects of treatment.
* History of major organ transplantation
* History of uncontrolled severe seizure disorder
* Inability to give informed written consent
* Serum creatinine > 1.5 x upper limit of normal
* AST and ALT > 2 x upper limit of normal
* Total bilirubin > 1.5 mg/ml
* No detectable PNH (paroxysmal nocturnal hemoglobinuria) clone where tested
* Concurrent hormonal contraceptive use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the ability of Pegylated Interferon Alfa-2a to achieve Complete Response or Partial Response in patients with (1) high risk polycythemia vera or (2) high risk essential thrombocythemia or (3) splanchnic vein thrombosis | 4 years

SECONDARY OUTCOMES:
To evaluate the toxicity and tolerability of therapy Pegylated Interferon Alfa-2a in each of the 3 strata by recording the number of adverse events that occur during the study by using CTC 4.0 as the guide. | 4 years
To measure the impact of Pegylated Interferon Alfa-2a on key biomarkers of the disease(s)by measuring the JAK2 allele burden. | 4 years
To evaluate specific pre-defined toxicity and tolerance of Pegylated Interferon Alfa-2a through a sequential structured symptom assessment package of patient reported outcome instruments. | 4 years
  Improvement in disease symptoms will be measured by the Myeloproliferative Neoplasm Symptom Assessment Form (MPN-SAF) instrument being used in this study.
To estimate survival, and incidence of development of myelodysplastic syndrome, myelofibrosis, or leukemic transformation during therapy Pegylated Interferon Alfa-2a. | 4 years
  We plan to capture the rate of disease progression to a more advanced myeloid malignancy.
Estimate the observed incidence of major cardiovascular events during therapy Pegylated Interferon Alfa-2a. | 4 years
  Capture and record the cardiovascular events that occur during the study.
To measure the impact of Pegylated Interferon Alfa-2a on JAK2-V617F, CALR, hematopoietic cell clonality in platelets and granulocytes in females, bone marrow histopathology, and cytogenetic abnormalities. | 4 years
  The impact of PEGASYS on JAK2 will be measured by the allele burden; hematopoietic cell clonality will be measured by whether patients with clonal disease return to polyclonal; bone marrow histopathology will be measured by going from abnormal to normal; cytogenetic abnormalities will be measured by seeing if the cytogenetics go from abnormal to normal.

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Ellen Ritchie, MD, Principal Investigator — Myeloproliferative Disorders-Research Consortium; Alessandro Rambaldi, MD, Principal Investigator — Myeloproliferative Disorders-Research Consortium
Locations (21):
- United States (16):
  - Mayo Clinic, Scottsdale, Arizona
  - The Palo Alto Clinic, Palo Alto, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Emory Hospital, Atlanta, Georgia
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Maryland, Baltimore, Maryland
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Geisinger Cancer Center, Danville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Italy (5):
  - Ospedale Riuniti de Bergamo, Bergamo, Italy
  - University Of Florence, Florence, Italy
  - Ospedale San Maartino Genova, Genova, Italy
  - San Matteo Hospital, Pavia, Italy
  - Universita Cattolica del Sacro Cuore, Rome, Italy

REFERENCES:
- [Derived] Thanarajasingam G, Bhatnagar V, Noble BN, Chen TY, Fiero MH, Hoffman R, Jeffery M, Mazza GL, Mascarenhas J, Mesa R, Murugappan M, Ross J, Sidana S, Warsame R, Kluetz PG, Dueck AC. Longitudinal graphics of patient-reported physical function in patients treated for hematologic malignancies. BMC Med Res Methodol. 2025 Aug 7;25(1):189. doi: 10.1186/s12874-025-02617-y. PMID 40775758